CLINICAL TRIAL: NCT02788474
Title: A 12-week, Double Blind, Randomised, Placebo Controlled, Parallel Group Trial Followed by a Single Active Arm Phase of 40 Weeks Evaluating the Effect of Oral Nintedanib 150 mg Twice Daily on Change in Biomarkers of Extracellular Matrix (ECM) Turnover in Patients With Idiopathic Pulmonary Fibrosis (IPF) and Limited Forced Vital Capacity (FVC) Impairment.
Brief Title: Effect of Nintedanib on Biomarkers of Extracellular Matrix Turnover in Patients With Idiopathic Pulmonary Fibrosis and Limited Forced Vital Capacity Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.227; 2015-003148-38 (EudraCT Number)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- nintedanib (Experimental)
  Interventions: Drug: nintedanib

INTERVENTIONS:
Drug: nintedanib
  Arms: nintedanib
Drug: placebo
  Arms: placebo

SUMMARY:
Identifying biomarkers to predict the clinical course and benefits of therapy early in the course of the disease remains one of the most urgent and relevant challenges to improve overall patient management, to prevent treatment delay or overtreatment. This study is conducted to examine the effect of nintedanib treatment on change in biomarkers indicative of extracellular matrix turnover which have been shown recently to correlate with disease progression. This study further aims to confirm the association of biomarker course during the first three months of treatment and disease progression.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent consistent with International Conference on Harmonisation Good Clinical Practice and local laws, signed prior to participation in the trial including any study related procedures being performed;
* Male or female patients aged >=40 years at Visit 1;
* A clinical diagnosis of Idiopathic pulmonary fibrosis (IPF) within the last 3 years from visit 0, based upon the American Thoracic Society/ European Respiratory Society /Japanese Respiratory Society/ Latin American Thoracic Association 2011 guideline;
* Chest high resolution computed tomography (HRCT) scan performed within 18 months of Visit 0;
* Combination of HRCT pattern, and surgical lung biopsy pattern (the latter if available) as assessed by central review are consistent with the diagnosis of Idiopathic pulmonary fibrosis;
* Forced vital capacity (FVC) >=80% of predicted normal at Visit 1.

Exclusion criteria:

* Alanine transaminase, Aspartate aminotransferase > 1.5 fold upper limit of normal (ULN) at Visit 1;
* Total bilirubin > 1.5 fold ULN at Visit 1;
* Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment);
* Relevant airways obstruction, i.e. pre-bronchodilator Forced expiratory volume in 1 second / Forced vital capacity < 0.70;
* History of myocardial infarction within 6 months of visit 1 or unstable angina within 1 month of Visit 1;
* Bleeding Risk:

  * Known genetic predisposition to bleeding;
  * Patients who require fibrinolysis, full-dose therapeutic anticoagulation or high dose antiplatelet therapy;
  * History of haemorrhagic central nervous system (CNS) event within 12 months prior to Visit 1;
  * History of haemoptysis or haematuria, active gastro-intestinal bleeding or ulcers and/or major injury or surgery within 3 months prior to Visit 1;
  * International normalised ratio (INR) > 2 at Visit 1;
  * Prothrombin time (PT) and partial thromboplastin time (PTT) > 150% of ULN at Visit 1;
* Planned major surgery during the trial participation, including lung transplantation, major abdominal or major intestinal surgery;
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of Visit 1;
* Creatinine clearance < 30 mL/min calculated by Cockcroft-Gault formula at Visit 1;
* Treatment with nintedanib, pirfenidone, azathioprine, cyclophosphamide, cyclosporine, any other investigational drug, n-acetylcysteine, prednisone/prednisolone >15 mg daily or >30 mg every 2 days OR use of other systemic corticosteroids as well as any investigational drugs within 4 weeks of Visit 2;
* Known hypersensitivity to nintedanib, peanut, soya or to any other components of the study medication;
* Prior discontinuation of nintedanib treatment due to intolerability/ adverse events considered drug related;
* A disease or condition which in the opinion of the investigator may interfere with testing procedures or put the patient at risk when participating in this trial;
* Alcohol or drug abuse which in the opinion of the treating physician would interfere with the treatment and would affect patient's ability to participate in this trial;
* Patients not able to understand and follow any study procedures such as but not limited to home spirometry, including completion of self-administered questionnaires without help;
* Women who are pregnant, nursing, who plan to become pregnant while in the trial or female patients with positive pregnancy (ß-HCG) test at Visit 1 and/or Visit 2;
* Women of childbearing potential4 not willing or able to use highly effective methods of birth control per International Conference on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Patients with acute IPF exacerbation or any respiratory tract infection in the four weeks prior to Visit 1 or during the screening period;
* Patients who are or have been participating in another trial with investigational drug/s within one month prior to Visit 1 and patients who have previously been enrolled in this trial;
* Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (86):
- United States (8):
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Western Connecticut Medical Group, Danbury, Connecticut
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Minnesota Lung Center, Minneapolis, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Clinical Research Solutions, Dayton, Ohio
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, Sydney, New South Wales
  - Concord General Repatriation Hospital -Ambulatory Care Unit, Concord, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (5):
  - ULB Hopital Erasme, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Czechia (5):
  - University Hospital Olomouc, Olomouc
  - University Hospital Plzen, Plzen-Bory, Pilsen
  - Thomayer Hospital, Prague
  - University Hospital Na Bulovce, Prague, Prague
  - Masaryk Hospital, Usti nad Labem, Ústí nad Labem
- Finland (5):
  - HYKS Keuhkosairauksien, Helsinki
  - KYS, Keuhkosairauksien, Kuopio
  - OYS, sisätautien klinikka, Oulu
  - Tampere University Hospital, Tampere
  - TYKS, Keuhkosairauksien klinikka, Turku, Turku
- France (7):
  - HOP de la Cavale Blanche, Brest
  - HOP Louis Pradel, Bron
  - HOP Européen G. Pompidou, Paris
  - HOP Maison Blanche, Reims
  - HOP Pontchaillou, Rennes
  - HOP Civil, Strasbourg
  - HOP Bretonneau, Tours
- Germany (10):
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Helios Klinikum Emil von Behring, Berlin
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsmedizin Greifswald, Greifswald
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum der Universität München - Campus Großhadern, München
  - Universitätsklinikum Münster, Münster
- Hungary (4):
  - Semmelweis University, Budapest
  - Csongrad County's Hosp., Deszk
  - Pulmonology Institute of Veszprem County, Farkasgyepu, Farkasgyepű
  - BAZ County Central Hospital and University Teaching Hospital, Miskolc
- Japan (10):
  - Tosei General Hospital, Aichi, Seto
  - Kurume University Hospital, Fukuoka, Kurume
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Kindai University Hospital, Osaka, Osakasayama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Tokushima University Hospital, Tokushima, Tokushima
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Global Health and Medicine Ctr, Tokyo, Shinjuku-ku
- Poland (6):
  - Our Doctor Clinical Trial Center, Department in Bydgoszcz, Bydgoszcz
  - Non-pub.Health Care NZOZ Profilaktyka W. Pierzchala,Katowice, Katowice
  - Univ. Hospital in Krakow,Pulmonology Clinical Dept, Krakow
  - John Paul II Cracovian Hosp, Krakow
  - Norbert Barlicki University Clinical Hospital No.1, Lodz, Lodz
  - Practice of Internists "Nasz Lekarz", Torun, Torun
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (13):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital de Galdakao, Galdakao
  - Hospital de Bellvitge, L'Hospitalet Llobregat (bcn)
  - Hospital La Princesa, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Puerta de Hierro, Majadahonda (Madrid)
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - CS Parc Taulí, Sabadell
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico de Valencia, Valencia
  - Hospital Dr. Peset, Valencia
- United Kingdom (6):
  - Southmead Hospital, Bristol
  - Papworth Hospital, Cambridge
  - Royal Devon and Exeter Hospital, Exeter
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Glaspole I, Bonella F, Bargagli E, Glassberg MK, Caro F, Stansen W, Quaresma M, Orsatti L, Bendstrup E. Efficacy and safety of nintedanib in patients with idiopathic pulmonary fibrosis who are elderly or have comorbidities. Respir Res. 2021 Apr 26;22(1):125. doi: 10.1186/s12931-021-01695-y. PMID 33902584
- [Derived] Noth I, Cottin V, Chaudhuri N, Corte TJ, Johannson KA, Wijsenbeek M, Jouneau S, Michael A, Quaresma M, Rohr KB, Russell AM, Stowasser S, Maher TM; INMARK trial investigators. Home spirometry in patients with idiopathic pulmonary fibrosis: data from the INMARK trial. Eur Respir J. 2021 Jul 8;58(1):2001518. doi: 10.1183/13993003.01518-2020. Print 2021 Jul. PMID 33419890
- [Derived] Maher TM, Stowasser S, Nishioka Y, White ES, Cottin V, Noth I, Selman M, Rohr KB, Michael A, Ittrich C, Diefenbach C, Jenkins RG; INMARK trial investigators. Biomarkers of extracellular matrix turnover in patients with idiopathic pulmonary fibrosis given nintedanib (INMARK study): a randomised, placebo-controlled study. Lancet Respir Med. 2019 Sep;7(9):771-779. doi: 10.1016/S2213-2600(19)30255-3. Epub 2019 Jul 17. PMID 31326319
- [Derived] Maher TM, Stowasser S, Nishioka Y, White ES, Cottin V, Noth I, Selman M, Blahova Z, Wachtlin D, Diefenbach C, Jenkins RG. Investigating the effects of nintedanib on biomarkers of extracellular matrix turnover in patients with IPF: design of the randomised placebo-controlled INMARK(R)trial. BMJ Open Respir Res. 2018 Aug 20;5(1):e000325. doi: 10.1136/bmjresp-2018-000325. eCollection 2018. PMID 30167310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial comprised of 2 treatment periods (52 weeks). The first treatment period was a 12-week, randomised, double-blind, placebo-controlled, parallel-group period whereas the second treatment period was a 40-week, single-arm, open-label, active treatment (nintedanib 150 milligram (mg) twice daily (bid)) period.
Pre-assignment Details: Participants with idiopathic pulmonary fibrosis (IPF) were eligible for the trial if they fulfilled all of the inclusion criteria and none of the exclusion criteria.
Groups:
- Placebo/ Nintedanib: Participants received soft gelatin capsules of matching placebo for 12 weeks in double blind period and Nintedanib 150 milligram (mg) twice daily (bid) for 40 weeks in open label period.
  1 capsule of Nintedanib 150 mg bid had possibility to be reduced to 100 mg bid to manage adverse events (AEs)
- Nintedanib/ Nintedanib: Participants received soft gelatin capsules of Nintedanib 150 mg bid for 12 weeks in double blind period and for 40 weeks in open label period.
  1 capsule of 150 mg bid had possibility to be reduced to 100 mg bid to manage adverse events (AEs)
Period: Double Blind Treatment Period
Arm/Group | Placebo/ Nintedanib | Nintedanib/ Nintedanib
Started (Randomised) | 231 | 116
Treated | 230 | 116
Completed | 221 | 112
Not Completed | 10 | 4
Not completed — Not treated | 1 | 0
Not completed — Patient's refusal | 3 | 0
Not completed — Adverse Event | 6 | 4
Period: Open Label Treatment Period
Arm/Group | Placebo/ Nintedanib | Nintedanib/ Nintedanib
Started | 221 | 112
Completed | 189 | 100
Not Completed | 32 | 12
Not completed — Adverse Event | 29 | 9
Not completed — Other than reason specified | 1 | 0
Not completed — Patient's refusal | 1 | 3
Not completed — Non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS), consisting of participants who were randomised to a treatment group and received at least one dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/ Nintedanib | Nintedanib/ Nintedanib | Total
Number analyzed (Participants) | 230 | 116 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.2) | 70.5 (7.7) | 70.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 23 | 84
  Male | 169 | 93 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Unreported data: Data not collected at sites in France due to local regulation
  Participants
    Hispanic or Latino | 19 | 9 | 28
    Not Hispanic or Latino | 193 | 96 | 289
    Unknown or Not Reported | 18 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants] — Unreported data: Data not collected at sites in France due to local regulation
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 68 | 35 | 103
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 144 | 70 | 214
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 18 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Change (Slope) in Blood C-reactive Protein Degraded by Matrix Metalloproteinase-1/8 (CRPM) From Baseline to Week 12.
Description: The rate of change (slope) in blood C-reactive protein degraded by matrix metalloproteinase-1/8 (CRPM) from baseline to week 12 is presented. The mean presented is the adjusted rate based on a random coefficient regression (CRPM log 10 transformed) with fixed effects for gender, age, height and random effect of patient specific intercept and time.
Time Frame: baseline and 12 weeks
Population: Treated set (TS) including participants with available data for this endpoint.
Measure: Mean (Standard Error); unit: nanogram/ millitre/ month (ng/ mL/ mth)
Arm/Group | Placebo/ Nintedanib | Nintedanib/ Nintedanib
Number analyzed (Participants) | 229 | 116
nanogram/ millitre/ month (ng/ mL/ mth) | -0.00190 (0.00165) | -0.00257 (0.00232)
Statistical Analysis 1: Comparison: Placebo/ Nintedanib vs Nintedanib/ Nintedanib; The rate of change (slope) in blood CRPM was assumed to be linear in each subject over the 12 weeks of treatment. The intercepts and slopes were assumed to be normally distributed with arbitrary covariance matrix. Since the distribution of the data was not normal, a log10 transformation was performed before conducting the statistical analyses. Significance tests were based on least-square means using 2-sided 95% confidence intervals (2-sided α=0.05); Test type: Other; p = 0.8146, random coefficient regression — random coefficient regression (random slopes and intercepts) model including sex, age and height as covariates (Due to the low number of measurements per patient, baseline CRPM was included as a response rather than as a covariate in the analysis); The Kenward-Roger approximation was used to estimate denominators degrees of freedom; Adjusted mean difference = -0.00066, 95% CI 2-sided [-0.00621 to 0.00488], Standard Error of Mean 0.00282 — Difference calculated as Nintedanib minus Placebo

2. Secondary Outcome: Percentage of Patients With Disease Progression as Defined by Absolute Forced Vital Capacity (FVC) Decline >=10% or Death Until Week 52
Description: For this endpoint, disease progression was defined by absolute FVC (percentage of predicted) decline ≥10% or death up to Week 52 based on in-clinic supervised spirometry.
  This is a key secondary endpoint of the trial. This outcome measure is "percentage of patients with disease progression" and CRPM is included in the various models as a factor/covariate, and that this outcome measure, the percentage of progressors are displayed under "Measured values"
Time Frame: 52 weeks
Population: Treated set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo/ Nintedanib | Nintedanib/ Nintedanib
Number analyzed (Participants) | 230 | 116
Percentage of participants | 30.43 [24.85 to 36.66] | 25.00 [18.01 to 33.60]
Statistical Analysis 1: Comparison: Placebo/ Nintedanib; To assess the association between disease progression (as defined by absolute forced vital capacity (FVC) decline >=10% or death) and the change in the Extracellular matrix (ECM) biomarker CRPM in the first 12 weeks, a logistic regression analysis including baseline blood CRPM and the monthly rate of change (slope) in blood CRPM in the first 12 weeks as covariates was applied for placebo-treated patients only to evaluate the potential of CRPM as a prognostic biomarker; Test type: Other; p = 0.2084, Regression, Logistic; slope estimate = 22.001, 95% CI 2-sided [-11.83 to 57.58] — Slope estimate is the monthly rate of change in CRPM up to week 12
Statistical Analysis 2: Comparison: Placebo/ Nintedanib vs Nintedanib/ Nintedanib; To assess how nintedanib treatment affected the association between disease progression (as defined by absolute forced vital capacity (FVC) decline >=10% or death) and the change in CRPM in the first 12 weeks, a logistic regression analysis including baseline blood CRPM, the monthly rate of change (slope) in blood CRPM up to Week 12, treatment and treatment-CRPM slope interaction as covariates was applied; Test type: Other; p = 0.1537, Regression, Logistic; slope estimate = -45.566, 95% CI 2-sided [-109.55 to 16.37] — Slope estimate is the monthly rate of change in CRPM up to week 12
Statistical Analysis 3: Comparison: Placebo/ Nintedanib vs Nintedanib/ Nintedanib; To assess whether the overall treatment regimen affected disease progression (as defined by absolute forced vital capacity (FVC) decline >=10% or death), a logistic regression analysis including baseline blood CRPM and randomised treatment as covariates was applied; Test type: Other; p = 0.3116, Regression, Logistic; Odds Ratio (OR) = 0.769, 95% CI 2-sided [0.46 to 1.27]
Statistical Analysis 4: Comparison: Placebo/ Nintedanib vs Nintedanib/ Nintedanib; To assess whether the monthly rate of change (slope) in blood CRPM in the first 12 weeks could explain the effect of treatment on disease progression (as defined by absolute forced vital capacity (FVC) decline >=10% or death), a logistic regression analysis including baseline blood CRPM, the rate of change (slope) in blood CRPM in the first 12 weeks and randomised treatment as covariates was applied; Test type: Other; p = 0.3175, Regression, Logistic; Odds Ratio (OR) = 0.772, 95% CI 2-sided [0.46 to 1.27]

3. Secondary Outcome: The Rate of Change in Blood Collagen 1 Degraded by Matrix Metalloproteinase-2/9/13 (C1M) From Baseline to Week 12
Description: The rate of change in blood Collagen 1 degraded by matrix metalloproteinase-2/9/13 (C1M) from baseline to week 12 is presented.
  The mean presented is the adjusted rate based on a random coefficient regression (C1M (negative reciprocal root transformation)) with fixed effects for gender, age, height and random effect of patient specific intercept and time.
Time Frame: baseline and 12 weeks
Population: Treated set (TS) including participants with available data for this endpoint.
Measure: Mean (Standard Error); unit: ng/ml/mth
Arm/Group | Placebo/ Nintedanib | Nintedanib/ Nintedanib
Number analyzed (Participants) | 229 | 116
ng/ml/mth | 0.00041 (0.00127) | 0.00162 (0.00172)
Statistical Analysis 1: Comparison: Placebo/ Nintedanib vs Nintedanib/ Nintedanib; The rate of change (slope) in blood C1M was assumed to be linear in each subject over the 12 weeks of treatment. Within-patient errors are modelled by an Unstructured variance-covariance matrix; Test type: Other; p = 0.5469, random coefficient regression — random coefficient regression model (C1M (negative reciprocal root-transformed)) with fixed effects for gender, age, height and random effect of patient specific intercept and time; Adjusted mean difference = 0.00121, 95% CI 2-sided [-0.00273 to 0.00515], Standard Error of Mean 0.00200 — Difference calculated as Nintedanib minus Placebo. Inter-individual variability is modelled by a Variance-Components variance-covariance matrix

4. Secondary Outcome: The Rate of Change in Blood Collagen 3 Degraded by Matrix Metalloproteinase-9 (C3M) From Baseline to Week 12
Description: The rate of change in blood Collagen 3 degraded by matrix metalloproteinase-9 (C3M) from baseline to week 12 is presented.
  The mean presented is the adjusted rate based on a random coefficient regression (C3M- log 10 transformation) with fixed effects for gender, age, height and random effect of patient specific intercept and time.
Time Frame: baseline and 12 weeks
Population: Treated set (TS) including participants with available data for this endpoint.
Measure: Mean (Standard Error); unit: ng/ml/mth
Arm/Group | Placebo/ Nintedanib | Nintedanib/ Nintedanib
Number analyzed (Participants) | 229 | 116
ng/ml/mth | -0.00091 (0.00158) | -0.00398 (0.00219)
Statistical Analysis 1: Comparison: Placebo/ Nintedanib vs Nintedanib/ Nintedanib; The rate of change (slope) in blood C3M was assumed to be linear in each subject over the 12 weeks of treatment. Within-patient errors are modelled by an Unstructured variance-covariance matrix; Test type: Other; p = 0.2429, random coefficient regression — random coefficient regression model (C3M (log10-transformed)) with fixed effects for gender, age, height and random effect of patient specific intercept and time; Adjusted mean difference = -0.00307, 95% CI 2-sided [-0.00823 to 0.00209], Standard Error of Mean 0.00262 — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious Adverse Event (SAE) & Non SAE: All adverse events (AEs) that occurred between first drug intake and 28 days after last drug intake (end of the Residual effect period (REP)); up to 53 weeks All cause mortality: All AEs during the course of the clinical trial; up to 56 weeks
Description: Treated set is used for reporting adverse events
Groups:
- Placebo (Double Blind Period): Participants received soft gelatin capsules of matching placebo for 12 weeks in double blind period.
- Nintedanib (Double Blind Period): Participants received soft gelatin capsules of Nintedanib 150 mg bid for 12 weeks in double blind period.
- Nintedanib (Open Label Period): Participants received soft gelatin capsules of Nintedanib 150 mg bid for 40 weeks in open label period. 1 capsule of 150 mg bid had possibility to be reduced to 100 mg bid to manage adverse events. Participants initially on placebo in the double blind period also received Nintedanib 150 mg bid in the open label period.
Arm/Group | Placebo (Double Blind Period) | Nintedanib (Double Blind Period) | Nintedanib (Open Label Period)
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/116 | 9/333
Serious Adverse Events (participants affected / at risk) | 18/230 | 8/116 | 65/333
Other Adverse Events (participants affected / at risk) | 103/230 | 80/116 | 277/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double Blind Period) (N=230) | Nintedanib (Double Blind Period) (N=116) | Nintedanib (Open Label Period) (N=333)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Pulmonary arteriovenous fistula (Congenital, familial and genetic disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 1 | 2
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2
Death (General disorders) | 0 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 1
Incarcerated hernia (General disorders) | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 5
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Influenza B virus test positive (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 2 | 1 | 1
Microscopic polyangiitis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double Blind Period) (N=230) | Nintedanib (Double Blind Period) (N=116) | Nintedanib (Open Label Period) (N=333)
Abdominal pain (Gastrointestinal disorders) | 8 | 6 | 16
Constipation (Gastrointestinal disorders) | 3 | 6 | 14
Diarrhoea (Gastrointestinal disorders) | 42 | 54 | 215
Nausea (Gastrointestinal disorders) | 15 | 17 | 57
Vomiting (Gastrointestinal disorders) | 7 | 9 | 42
Bronchitis (Infections and infestations) | 5 | 3 | 23
Lower respiratory tract infection (Infections and infestations) | 7 | 4 | 18
Nasopharyngitis (Infections and infestations) | 19 | 10 | 49
Upper respiratory tract infection (Infections and infestations) | 9 | 3 | 20
Alanine aminotransferase increased (Investigations) | 2 | 7 | 17
Aspartate aminotransferase increased (Investigations) | 4 | 6 | 16
Gamma-glutamyltransferase increased (Investigations) | 2 | 5 | 17
Weight decreased (Investigations) | 2 | 6 | 26
Decreased appetite (Metabolism and nutrition disorders) | 10 | 12 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 24
Headache (Nervous system disorders) | 7 | 7 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 5 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT02788474/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT02788474/SAP_001.pdf